CLINICAL TRIAL: NCT03729154
Title: Preschool First Step to Success: An Efficacy Replication Study
Acronym: PFS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R32 4A150221
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Oppositional Defiant Disorder
MeSH Terms: conditions — Oppositional Defiant Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Step (Experimental): First Step is a comprehensive early intervention that is delivered by a behavioral coach who works in collaboration with the classroom teacher and parents. First Step addresses moderate to severe behavior problems of young children and includes both classroom and home components. The program takes about three months from start to finish and requires approximately 60 hours of the coach's time for implementation over this three month period.
  Interventions: Behavioral: First Step
- Treatment as Usual (No Intervention): Participants in the Treatment as Usual condition will receive behavioral and counseling services typically provided by their preschool.

INTERVENTIONS:
Behavioral: First Step — First Step is a comprehensive early intervention that is delivered by a behavioral coach who works in collaboration with the classroom teacher and parents. First Step addresses moderate to severe behavior problems of young children and includes both classroom and home components. The program takes about three months from start to finish and requires approximately 60 hours of the coach's time for implementation over this three month period.
  Arms: First Step

SUMMARY:
The purpose of this research is to conduct a Goal 3 efficacy study to replicate the positive effects of the preschool version of the First Step intervention- Preschool First Step (PFS)-in improving social/behavioral and academic outcomes to support learning, and to begin to identify the utility of the intervention (i.e., the degree to which it is feasible and practical for implementation in authentic school settings). The primary goal is to replicate the impressive FS outcomes previously reported. The second goal is to mantle the PFS intervention for dissemination at the program-rather than the classroom-level by addressing several aspects of implementation and sustainability in preparation for a Goal 4 (Effectiveness) trial. PFS was developed via a 5-year Head Start University Partnership grant from the Administration for Children, Youth, and Families to adapt FS for Head Start populations.

DETAILED DESCRIPTION:
Children with conduct and oppositional defiant disorders require a substantial effort for remediation. Longitudinal research indicates that increased antisocial behavior and impairments in social competence skills often serve as harbingers of future adjustment problems in a number of domains including mental health, employment, and academic achievement. It is critical to divert at-risk children from this path as soon as possible in their lives and school careers through early, coordinated interventions involving parents and caregivers, teachers and peers. Preschool is an ideal setting for accomplishing this task in collaboration with families.

The purpose of this project is to conduct a Goal 3 efficacy study to replicate the positive effects of the preschool version of the First Step to Success intervention in improving social/behavioral and academic outcomes to support learning, and to begin to identify the utility of the intervention (i.e., the degree to which it is feasible and practical for implementation in authentic school settings). Ideally, this project will result in an intervention option for serving young children with severely challenging behavior across home and school settings that meets the What Works Clearinghouse evidence standards. The preschool version of First Step is a fully developed, manualized intervention that targets social emotional and academic outcomes for young children with severe behavior problems. This application outlines a 4-year randomized efficacy trial in which the primary goal is to replicate the impressive outcomes previously reported. The second goal is to mantle the First Step intervention for dissemination at the program- rather than the classroom-level by addressing several aspects of implementation and sustainability in preparation for a Goal 4 (Effectiveness) trial. Results from a nearly completed NICHD-funded efficacy trial (R01HD055334) provide promising evidence that exposure to the intervention reduced participating children's problem behaviors and increased children's social skills. Further, the available evidence suggests that the preschool version of First Step can be implemented with fidelity, and that the intervention procedures are acceptable to coaches, parents, and teachers in preschool settings.

For this application, preschool programs (Head Start) serving a diverse group of low income families in rural and urban Oregon and Kentucky have all agreed to participate in this study. This Goal 3 efficacy-replication research application strategically prepares for a future effectiveness study with (a) efficacy supported by at least two rigorous trials, (b) specific intervention enhancements for training and supervision and (c) measurement and design to test efficacy at a broader site/building level rather than classroom. Pre, post, follow-up and one-year follow-up data will be collected. Measures to be included in this proposed research are questionnaire measures completed by parents and/or teachers, direct assessment of the child's academic level (school readiness), direct observations of the classroom environment, and implementation and process measures of treatment integrity. The study will utilize a cluster randomized controlled trial design that nests teachers and classrooms within early childhood buildings/sites. Project staff will recruit 48 EC sites/buildings (24 in Kentucky and 24 in Oregon) having 192 low-income families with preschoolers that meet inclusion criteria and agree to participate in the study and, after completion of screening procedures and baseline data collection, will use a matched pair randomization procedure to assign 24 to a Preschool First Step intervention condition and 24 to a business-as-usual control condition. Investigators will utilize the mixed-model ANCOVA approach when examining differences between intervention and control groups on outcomes, process and social validity measures. Results from this replication study will provide the fields of general and special education with (a) important evidence that First Step is reliably effective in reducing problem behaviors and increasing the prosocial behavior repertoire of preschool children and (b) an exploratory investigation of contextual factors that are important for implementation success.

ELIGIBILITY:
Inclusion Criteria:

*Children at-risk for development of Oppositional Defiant Disorder with high scores exceeding normative criteria on the Systematic Screening for Behavior Disorders (Walker, Severson, & Feil, 2014).

Exclusion Criteria:

*Children with significant psychopathology, such as schizophrenia.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Social Skills Improvement System Rating Scale | Change from Baseline Social Skill Score at 4 months, 8 months, 12 months and 16 months
  The Social Skills Improvement System Rating Scale(Gresham & Elliot, 2008) is the second edition of the Social Skills Rating System and provides a measure of peer-to-peer and teacher-related social skills. The Social Skills subscale of the SSiS-RS is a rating scale completed by teachers and parents across the social skill domain on a 4-point scale from 0=Never, 1= Seldom, 2=Often to 3=Almost Always,
Change in Problem Behavior Scale | Change from Baseline Problem Behavior Score at 4 months, 8 months, 12 months and 16 months
  The Problem Behavior Scale from the Social Skills Improvement System Rating Scale (Gresham & Elliot, 2008) is the second edition of the Social Skills Rating System. The Problem Behavior Scale is a rating scales completed by teachers and parents across problem behavior domain on a 4-point scale from 0=Never, 1= Seldom, 2=Often to 3=Almost Always,
Change in Teacher-Student Conflict | Change from Baseline Problem Behavior Score at 4 months, 8 months, 12 months and 16 months
  The Teacher-Student Conflict instrument provides a measure of child-to-teacher relationship. The Teacher-Student is a rating scale completed by teachers regarding their interactions with the participating child, such as "Dealing with this child drains my energy" and "Despite my best efforts, I'm uncomfortable with how this child and I get along" on a 5-point scale from 0=Definitely does not apply, 1=Does not really apply, 2=Neutral, not sure, 3=Applies somewhat to 4=Definitely applies.

CONTACTS AND LOCATIONS:
Overall Officials: Edward G Feil, Ph.D., Principal Investigator — Oregon Research Institute